CLINICAL TRIAL: NCT06618443
Title: Effect of Scapular Mobilization With Arm Movement on Shoulder Pain and Range of Motion and Disability in Older Adults With Adhesive Capsulitis.
Brief Title: Scapular Mobilization With Arm Movement in Patients With Adhesive Capsulitis.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beni-Suef University (Other)
Responsible Party: Principal Investigator, Ayman Mohamed, Associate Professor, Beni-Suef University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BNS
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Shoulder Adhesive Capsulitis
Keywords: scapular mobilization; arm movement; pain; range of motion; disability; older adults; adhesive capsulitis
MeSH Terms: conditions — Bursitis; Pain | interventions — Movement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scapular mobilization with movement (Experimental): The treatment consisted of scapular mobilization with arm movement in all directions for 15 min/session for 3 sessions/week for 4 weeks. Scapular mobilization included scapular upward glide and downward glid. Scapular upward glide was performed with shoulder adduction and extension, while scapular downward glide was performed with shoulder abduction and flexion.
  Interventions: Other: Scapular mobilization with movement
- Control (No Intervention)

INTERVENTIONS:
Other: Scapular mobilization with movement — The treatment consisted of scapular mobilization with arm movement in all directions for 15 min/session for 3 sessions/week for 4 weeks. Scapular mobilization included scapular upward glide and downward glid. Scapular upward glide was performed with shoulder adduction and extension, while scapular downward glide was performed with shoulder abduction and flexion.
  Arms: Scapular mobilization with movement

SUMMARY:
50 patients with shoulder adhesive capsulitis were admitted. the patients will receive scapular mobilization (downward or upward mobilization) associated with arm movements. The percentage of improvement in shoulder ROM of flexion, abduction, and external rotation; and decrease in shoulder pain and disability index (SPADI).

ELIGIBILITY:
Inclusion Criteria:

* The existence of unilateral adhesive capsulitis (stage II) with incapability of the participant to raise the arm more than 100 degrees in the plane of the scapula

Exclusion Criteria:

* The presence of any shoulder problem contraindicated for performing exercises to the shoulder joint, such as active inflammatory disease, cancer, active infection, recent subluxations or dislocations, fractures, and surgeries near the shoulder region.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-02-15 (Estimated)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 3 months
  The patient was asked to refer to the degree of their shoulder problems in the previous week by choosing a number on a scale from 0 (no pain or disability) to 10 (extreme pain and disability) for each question 13. The chosen number from each subscale was summed up and transformed into an out-of-100 score. The mean two scales were assigned a sum score out of 100. The higher the end score, the more shoulder pain, or disability.
Shoulder range of motion of flexion, abduction, and external rotation | 3 months
  For evaluating shoulder flexion and abduction, the goniometer was positioned on the distal arm. The patient sat in a vertical position on an elevated-backed chair. To restrain trunk unwanted motion, a belt was put around the patient's waist and chair. The patient was directed to lift the tested arm voluntarily with his palm facing the floor.
  For evaluating shoulder external rotation, the goniometer was positioned on the proximal forearm next to the wrist joint. The patient was asked to lie supine with flexed hips and knees 45 degrees. The tested arm was placed on the plinth with 90 degrees in shoulder abduction, 90 degrees in elbow flexed, and 0 degrees in wrist joint11. The patient was asked to turn the forearm up to externally rotate the arm.
Scapular dyskinesis | 3 months
  this test was conducted with grasping dumbbells following the bodyweight, 1.4 kg (3 lb) for patients with a weight of lower than 68.1 kg (150 lb), and 2.3 kg (5 lb) for patients with a weight of 68.1 kg or higher. If any patient was unable to carry these predetermined weights, the weight was decreased by 0.5 kg29. Then, the patient was instructed to instantaneously raise his arms overhead with thumbs-up as much as possible at a 3-second count and then lower the arms back to the same starting position at a 3-second count.
  This study used a caliper to develop an objective method to measure improved scapular dyskinesis. The height difference between the 2 scapulae was measured with a caliper to the nearest millimeters at the end of the available shoulder ROM. The height difference between the 2 scapulae was defined as the difference between the vertical positions of the 2 inferior angles of the 2 scapulae30. A distance of more than 75 mm between the 2 scapulae was c
Electromyography | 3 months
  Electromyographical analysis of Upper and Lower trapezius and Serratus anterior

IPD SHARING:
Plan to Share IPD: Undecided